CLINICAL TRIAL: NCT02052219
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study to Evaluate the Efficacy and Safety of Blisibimod Administration in Subjects With IgA Nephropathy
Brief Title: BRILLIANT-SC: A Study of the Efficacy and Safety of Blisibimod Administration in Subjects With IgA Nephropathy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN-IGN3331
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: IgA Nephropathy
Keywords: Blisibimod; IgA nephropathy; BAFF; BLyS
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — AMG623 peptibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blisibimod (Experimental)
  Interventions: Drug: Blisibimod
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Blisibimod — Blisibimod administered subcutaneously
  Arms: Blisibimod
Drug: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effect of blisibimod plus standard of care versus placebo plus standard of care alone on the proportion of subjects achieving improvement in renal disease parameters.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Biopsy-proven IgA nephropathy
* Proteinuria ≥ 2g/24hr or equivalent
* Receiving physician-directed optimized standard of care that includes ACEI and/or ARB.
* Estimated glomerular filtration rate (eGFR) >40mL/min/1.73m2

Exclusion Criteria:

* Clinical or histologic evidence of non-IgA-related glomerulonephritis
* IgA nephropathy with greater than 50% glomerulosclerosis or cortical scarring
* Meets eGFR criteria
* Malignancy within past 5 years
* Known to be positive for HIV and/or positive at the screening visit for hepatitis B, or hepatitis C
* Liver disease
* Neutropenia
* Active infection requiring hospitalization or treatment with parenteral antibiotics within the past 60 days or history of repeated herpetic viral infections
* History of active tuberculosis or a history of tuberculosis infection
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects to achieve the proteinuria threshold | Week 24
The proportion of subjects who progress to end-stage renal disease | approximately 5 years

SECONDARY OUTCOMES:
Change from baseline in serum immunoglobulins IgA, IgG and IgM, plasma cells and B cell subsets | Week 24
Number of Participants with Adverse Events | Week 24
Change from baseline in serum creatinine | Week 24
Change from baseline in eGFR | Week 24
The proportion of subjects requiring the addition of corticosteroid or other therapy | Week 24